CLINICAL TRIAL: NCT03114098
Title: Personalized Medicine: Pharmacogenetics Anomaly Research in Children and Adolescents With Pharmacological Resistance to Psychotropic Drugs
Brief Title: Pharmacogenetics Anomaly Research in Children and Adolescents With Pharmacological Resistance to Psychotropic Drugs
Acronym: M4P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-HPNCL-02
Record Dates: First submitted 2017-02-22; First posted 2017-04-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-07

CONDITIONS: Drug Resistance; Psychotropic Drugs
Keywords: Drug Resistance; CYP2D6; cytochrom P450

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CYP2D6 gene abnormalities (Experimental): * A salivary sample (2 ml sample) which will allow the investigation of an anomaly of the metabolism of psychotropic drug.
  * Blood sampling will be performed to assess treatment tolerance (6 ml). A sample (4 ml) will be kept for possible future analyzes in relation to the objectives of this study for the recruiting center of Nice.
  * Electrocardiogram
  * Clinical exam
  * Clinical Global Impression Scale (CGI-S)
  * Children's Global Assessment Scale (CGAS)
  * Sheehan Disability Scale (SDS)
  * Wechsler Preschool and Primary Scale of Intelligence III (WPPSI-III )
  * Wechsler Intelligence Scale for Children - 4 (WISC-4)
  * Wechsler Adult Intelligence Scale 4 (WAIS 4)
  * Diagnostic and Statistical Manual of Mental Disorders (DSM)
  * Autism Diagnostic Interview (ADI)
  Interventions: Other: gene abnormalities

INTERVENTIONS:
Other: gene abnormalities — A salivary sample (2 ml sample) Blood sampling will be performed to assess treatment tolerance (6 ml)

SUMMARY:
Psychotropic drugs are frequently used in children and adolescents in France with a prescription rate of 2.5%. Antipsychotics (PA) and antidepressants (AD), each concern 0.3% of the pediatric population (Kovess et al., 2015). Despite appropriate pharmacological treatment, some patients are drug-resistant and have persisting symptoms and ineffective psychotropic treatments. These children and adolescents are generally exposed to many psychotropic molecules and often to poly-therapy.

Most psychotropic treatments, especially AP and AD, are metabolised at the hepatic level by cytochrome P450 and in particular by CYP2D6. Duplication / multiplication of the CYP2D6 gene induces too rapid metabolism of drugs.

Demonstration of a CYP2D6 abnormality has a direct impact on the management of the patient and on the clinical decisions of the clinician. Thus, knowledge of individual metabolism will decrease the failure of treatment, improve quality of life and therapeutic compliance.

DETAILED DESCRIPTION:
Psychotropic drugs are frequently used in children and adolescents in France with a prescription rate of 2.5%. Antipsychotics (PA) and antidepressants (AD) each concern 0.3% of the pediatric population (Kovess et al., 2015). Despite appropriate pharmacological treatment, some patients are drug-resistant and have persisting symptoms and ineffective psychotropic treatments. These children and adolescents are generally exposed to many psychotropic molecules and often to poly-therapy. Additionally, hospitalizations for child psychiatry, sometimes of prolonged duration, are frequent for these patients. In France, to date, the psychiatrist practitioner rarely uses pharmacogenetic evaluation as a complementary tool for prescribing psychotropic drugs. Nevertheless, an individualized prescription taking into consideration the patient's individual metabolism could greatly improve the benefit and reduce the risk of psychotropic treatments in the pediatric population.

Most psychotropic treatments, especially AP and AD, are metabolised at the hepatic level by cytochrome P450 and in particular by CYP2D6. Duplication / multiplication of the CYP2D6 gene induces too rapid metabolism of the drugs (ultrafast metabolizer). It is linked to a clinical inefficiency of treatments, and concerns up to 10% of the general population in southern Europe (Scordo et al., 2004).

In a preliminary study in Nice, an abnormality of CYP2D6 was found in 4 of the 7 patients tested with drug-resistant and / or with numerous adverse effects to the AP, of which 3 of the 5 pharmacologically resistant patients shows a duplication of the gene.

Demonstration of a CYP2D6 abnormality has a direct impact on the management of the patient and on the clinical decisions of the clinician. Thus, knowledge of individual metabolism will decrease the failure of treatment, improve quality of life and therapeutic compliance.

ELIGIBILITY:
Inclusion Criteria:

* Pharmaco resistance to psychotropic drugs
* Obtaining the informed consent of the patient and his / her parents or legal guardian
* Affiliation to a social security system

Exclusion Criteria:

* Patient deprived of liberty

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
prevalence of a CYP2D6 duplication or polymorphisms | At baseline
  study the prevalence of a CYP2D6 duplication or polymorphisms associated with an ultrafast metabolizing phenotype in a population of children and adolescents who are drug-resistant to antipsychotic and antidepressant psychotropic drugs. performed by analysis of salivar sample

SECONDARY OUTCOMES:
Psychiatric diagnosis and comorbidities | At baseline
  Diagnostic and Statistical Manual of Mental Disorders 5 DSM5
Global Severity of illness | At baseline
  Clinical Global Impression scale (échelle CGI-I)
Severity of illness for children | At baseline
  Children's Global Assessment Scale (CGAS)
Current and previous psychotropic treatment | At baseline
  Number of different molecules (antipsychotic antidepressant) used during the therapeutic history of the patient, duration of treatment with each molecule, type and maximum dose of current and previous psychotropic treatments.
Side effects in different psychotropic treatments | At baseline
  Type and severity of the adverse effects identified during the various psychotropic treatments will be collected. This collection will be carried out through the interrogation and study of the medical file
New anomalies of CYP2D6 gene | At baseline
  To look for any other abnormality of the CYP2D6 gene not known to be associated with an ultrafast metabolizing phenotype
Description of the clinical phenotype of patients | At baseline
  The characterization of the clinical phenotype will be carried out on the one hand by the standardized diagnostic interview MINI Mini International Neuropsychiatric Interview

CONTACTS AND LOCATIONS:
Overall Officials: Susanne THÜMMLER, MD, Principal Investigator — Fondation Lenval Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Fondation Lenval Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice, France

IPD SHARING:
Plan to Share IPD: No